CLINICAL TRIAL: NCT06787534
Title: The Favorable Impact of Hepatitis B Core Antibody Positive Grafts on Liver Transplantation for Hepatitis B Virus-related Hepatocellular Carcinoma: a Nationwide Multicenter Retrospective Cohort Study
Brief Title: The Favorable Impact of HBcAb Positive Grafts on Liver Transplantation for HBV-related HCC
Status: Completed | Type: Observational
Sponsor: Xiao Xu (Other)
Responsible Party: Sponsor-Investigator, Xiao Xu, Prof., Zhejiang University
Organization: Zhejiang University (Other)
Other Study IDs: CT-2025-ZJU-OBS01
Record Dates: First submitted 2025-01-14; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HBcAb negative group: Liver transplant recipients with HBcAb negative grafts
  Interventions: Other: No Interventions
- HBcAb positive group: Liver transplant recipients with HBcAb positive grafts
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions

SUMMARY:
The utilization of marginal grafts may help alleviate the demand mismatch. However, strategies to optimize the use of hepatitis B core antibody (HBcAb) positive grafts still requires further investigation. This study aims to investigate possible interactions between HBcAb positive grafts, HCC and HBV-related diseases, and long-term patient and graft survival. The study retrospectively analyzed patients undergoing liver transplantation in 8 centers between January 2015 and December 2020.

DETAILED DESCRIPTION:
This retrospective observational study included patients who underwent liver transplantation between January 2015 and December 2020 from 8 transplant centers in China, including the First Affiliated Hospital, Zhejiang University School of Medicine, Shulan (Hangzhou) Hospital, the Affiliated Hospital of Qingdao University, the Third Affiliated Hospital of Sun Yat-sen University, West China Hospital of Sichuan University, HuaShan Hospital of Fudan University, Beijing Chaoyang Hospital of Capital Medical University, and the Second Xiangya Hospital of Central South University. Demographic and clinicopathological data of these patients were extracted from the prospectively maintained China Liver Transplant Registry (CLTR) database. The exclusion criteria were as follows: (1) re-transplantation, combined organ transplantation or living donor liver transplantation; (2) intrahepatic cholangiocarcinoma or combined hepatocellular-cholangiocarcinoma; (3) HBsAg positive graft; and (4) missing of baseline data. Patients who were lost to follow-up were also excluded.

Statistical analysis was performed with GraphPad Prism (Version 9), IBM SPSS Statistics (Version 26) and R version 4.3.1 (R Foundation). Regarding the initial demographic data, continuous variables were depicted as medians (IQR: Inter-Quartile Range) and analyzed for differences with the Mann-Whitney U test. Categorical variables were contrasted through the application of the chi-squared test. Cumulative patient survival, graft survival, recurrence-free survival and recurrence rate were analyzed by the Kaplan-Meier method and compared with the log-rank test. To lessen the impact of potential confounders and selection bias, propensity score matching (PSM) was implemented to form comparable groups. Unbalanced variables were entered into the 1:1 matching model. Cox proportional hazard models were used to estimate hazard ratios (HRs) with 95% confidence intervals (CIs) for the relationship between variables and the event of interest. Univariate analyses were performed to identify the potential risk factors for patient survival, graft survival and recurrence-free survival in each group. Variables (P<0.10) were included in the backward stepwise multivariate analyses.

ELIGIBILITY:
Inclusion Criteria:

* (1) primary transplantation; (2) complete baseline data.

Exclusion Criteria:

* (1) re-transplantation, combined organ transplantation or living donor liver transplantation; (2) intrahepatic cholangiocarcinoma or combined hepatocellular-cholangiocarcinoma; (3) HBsAg positive graft; and (4) missing of baseline data. Patients who were lost to follow-up were also excluded.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Of the patients, 18.4% were female, and the median age of the patients was 50 years (range 18-82 years; IQR 43-56 years). The median value of the laboratory MELD score was 25 (IQR 13-35). The median follow-up duration for the study cohort was 44.7 months (IQR 16.0-65.3 months).
Sampling Method: Non-Probability Sample
Enrollment: 6924 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative death | 2015.1.1-2023.12.31
  The death of a patient following liver transplanation

SECONDARY OUTCOMES:
Postoperative recurrence | 2015.1.1-2023.12.31
  The day of hepatocellular carcinoma recurrence